CLINICAL TRIAL: NCT01857570
Title: Volume CT of the Wrist and Carpus After Trauma: A Pilot Study
Brief Title: Volume CT of the Wrist and Carpus After Trauma
Acronym: VuisT
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: NL43482.091.13
Record Dates: First submitted 2013-05-10; First posted 2013-05-20 (Estimated); Last update posted 2015-05-14 (Estimated); Status verified 2015-05

CONDITIONS: Wounds and Injuries; Wrist Injuries
Keywords: Radius fracture; Scaphoid fracture; Tomography, x-ray computed
MeSH Terms: conditions — Wounds and Injuries; Wrist Injuries; Radius Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adult, clinical suspicion fractures wrist or carpus: - Patients (18 years and older) who are referred to our hospital for conventional radiography of the wrist and carpus
  Interventions: Radiation: Volume Computed Tomography of the wrist and carpus

INTERVENTIONS:
Radiation: Volume Computed Tomography of the wrist and carpus

SUMMARY:
The purpose of this study is to evaluate whether standard volume computed tomography (CT) has impact on treatment in patients with suspicion of fractures of the wrist and carpus.

ELIGIBILITY:
Inclusion Criteria:

* Patients (18 years and older) who are referred to our hospital for conventional radiography of the wrist and carpus
* Recent trauma mechanism (within 3 days before presentation)
* Clinical suspicion of fractures of the wrist and carpus. The carpus includes all carpal bones, but does not include the metacarpal bones.

Exclusion Criteria:

* Patients who were not evaluated by a clinician before imaging was performed.
* Open fractures
* No informed consent or no prospective data collection could be obtained. Informed consent cannot be obtained in case patients do not speak or understand Dutch.
* Patients who cannot be positioned in upright position, immobilized on a spine board or transferred to the intensive care unit and cannot undergo upright CT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients who enter the emergency or radiology department of the Radboud University Nijmegen Medical Centre for suspicion on fractures of the wrist and study are eligible for this study.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2013-06; Primary Completion 2014-04 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with prospectively documented treatment changes after CT | within same visit (i.e. in one day)
  This endpoint is defined as presence of difference in predefined treatment regimens before and after CT. These regimens include:
  -Conservative treatment on the emergency ward (functional, immobilization with bandage, cast, or closed reduction and cast), closed operative treatment (reduction and cast on operation room, percutaneous pinning, or external fixation), open surgical treatment (dorsal, radial, or palmar exposure with reduction and internal fixation).
  Additional regimens include: Second opinion from a colleague or consulting a different specialism.

SECONDARY OUTCOMES:
Diagnostic performance of CT and conventional radiography (CR) for fracture pattern | within the same visit (one day)
  Fracture patterns are classified according to presence and type of fractured bones, presence of intra-articular components of distal radius fractures (including sigmoid notch involvement), presence of (fracture) dislocation or avulsion fractures of carpal bones. Standard of reference is presence of injuries at imaging, at surgery, and disability complains at 1-year follow up. In case of discrepancy, consensus will be reached at the end of the study by a panel of trauma surgeons and radiologists.

OTHER OUTCOMES:
Radiological feasibility | Within an average of three days after CT
  Image quality (5-point scale), artifacts (5-point scale) noise (standard deviation Hounsfield Units), radiation dose, and presence of technical problems
Patient outcome: Pain and disability | one year
  Pain and disability according to the "Patient rated wrist and hand evaluation (PRWHE) score" 6 weeks, 6 months, and 12 months after trauma

CONTACTS AND LOCATIONS:
Overall Officials: Mathias Prokop, MD, PhD, Principal Investigator — Radboud University Medical Center; Monique Brink, MD, PhD, Study Chair — Radboud University Medical Center
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Netherlands